CLINICAL TRIAL: NCT01808196
Title: A Preliminary, Open-label Trial of Losartan Potassium in Participants With Eosinophilic Esophagitis (EoE) With or Without a Connective Tissue Disorder.
Brief Title: Testing Effectiveness of Losartan in Patients With EoE With or Without a CTD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0106
Record Dates: First submitted 2013-01-30; First posted 2013-03-11 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-08

CONDITIONS: Eosinophilic Esophagitis; Connective Tissue Disorders
Keywords: Eosinophilic Esophagitis; Connective Tissue Disorders; Drug trial
MeSH Terms: conditions — Eosinophilic Esophagitis; Connective Tissue Diseases | interventions — Losartan; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: This study is an open-label study which means that all participants receive the study medicine
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Losartan (Experimental): Participants with eosinophilic esophagitis receive Losartan daily
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Losartan Potassium — The dose of study drug is dependent on body weight and tolerance but did not exceed 100 mg.
  Other Names: Angiotensin II Receptor Antagonists

SUMMARY:
The purpose of this research study is to test the safety of losartan potassium and see what effects (good and bad) it has on you and your eosinophilic esophagitis.

DETAILED DESCRIPTION:
Losartan is a drug that is approved by the United States Food and Drug Administration (FDA) for use in adults and children over 6 years of age who have high blood pressure. Losartan has been safe when administered to patients with normal blood pressure. This medication has not been studied in people with eosinophilic esophagitis or connective tissue disorder. Eosinophils are a type of white blood cell that induces inflammation. Eosinophils with other inflammatory cells produce a protein called TGF-β, which may contribute to part of EoE. Losartan may reduce the amount of this protein and therefore, be a treatment for eosinophilic esophagitis.

You will be in the research study for approximately 4 months. Participation in this research study will involve 9 study visits. Of the 9 study visits, at least 3 visits will take place in the clinic; the other visits may take place over the telephone.

Throughout the study, the following activities will occur:

1. A physical and vital signs will be obtained
2. There will be two endoscopies performed one at the beginning and one at the end of the study
3. Blood will be obtained up to three times
4. Pregnancy tests will be performed
5. Quality-of-life questionnaires will be completed

This is an open-label trial, which means that if you choose to enroll and you meet screening criteria, you will receive Losartan as a treatment. You will start the study drug at a low dose. It will be increased at vist 3 the 1 month visit. The dose of study drug will be increased depending on your weight and how well you tolerate each dose but will not exceed 100mg of study drug per day. It may be increased or decreased during the study if there are any side effects. If you do not have certain side effects, you will take each dose of the study drug between 21 and 28 days until your next study visit. You will swallow a pill or liquid once or twice a day.

This study will consist of 4 phases: screening, treatment (titration and maintenance), end of treatment, and follow-up. Participants that are between 5 to 18 years of age, as well as the parent or legal guardian will be asked to complete questionnaires of quality-of-life symptom severity questionnaires. Participants between the age of 19 and 21 will also have to fill out these questionnaires, but parents/guardians will not have to fill these out. If you are the parent or caretaker, the only study activity in which you will be involved is the completion of questionnaires about you and your family.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of eosinophilic esophagitis.
2. Have been on a high dose proton pump inhibitor for at least 8 weeks prior to a diagnostic endoscopy of eosinophilic esophagitis without histologic resolution.
3. Agree to maintain the same diet throughout the duration of the study.
4. If participant is female: meet one of the following criteria:

   1. Is of non-childbearing potential (pre-menarchal or surgically sterile with documentation)
   2. Is of childbearing potential with a negative urine pregnancy test at screening.

Exclusion Criteria:

1. Past or planned cardiac surgeries.
2. Had an aortic root Z-score greater than 3 on a previous echocardiogram.
3. Have intolerance to the study agent such as angioedema, IgE-mediated allergy.
4. Have renal dysfunction with creatinine in excess of the upper normal limit for age.
5. Have another disorder that causes esophageal eosinophilia (e.g., hypereosinophilic syndrome, Churg Strauss vasculitis, eosinophilic granuloma, or a parasitic infection).
6. Diagnosed with hepatic insufficiency.
7. History of abnormal gastric or duodenal biopsy or documented gastrointestinal (GI) disorders (e.g., Celiac Disease, Crohn's disease or helicobacter pylori infection.), not including chronic gastritis, chronic duodenitis, mucosal eosinophilia or other eosinophilic gastrointestinal disorders.
8. Used anti-immunoglobulin E [IgE] mAb, anti-tumor necrosis factor [TNF] mAb, anti-IL-5 agents, or anti-IL-13 within the last six months.
9. Used methotrexate, cyclosporine, interferon-α, or other systemic immunosuppressive or immunomodulating agents within the last three months.
10. Have a history of a stricture during an endoscopy procedure that prevents passage of the endoscope.
11. Taking or plan to take an angiotensin II receptor blocker (ARB) therapy, angiotensin-converting enzyme inhibitor (ACEI), beta blocker therapy (BB), or calcium channel blocker at the screening visit or at any time during the study, or have you been taking any of these medications for the last three months.
12. If the participant is female: pregnant or nursing.
13. Taking any investigative drug or device study within the last 30 days.
14. Had participated in any investigative biologics study within the last three months prior to the study entry.
15. Taking or plan to take hydrochlorothiazide, warfarin, cimetidine, phenobarbital, rifampin, or fluconazole.
16. If the participant is female: using a medically accepted effective method of birth control.
17. Will be able to complete all study procedures including endoscopy.
18. Taking or plan to take potassium supplements or salt substitutes containing potassium.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2015-01-13 (Actual); Study Completion 2015-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Pablo Abonia, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Marc E Rothenberg, M.D., Ph.D., Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Kara Kliewer, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan: Participants with eosinophilic esophagitis receive the Losartan daily
  Losartan Potassium: The dose of study drug is dependent on body weight and tolerance but did not exceed 100 mg.
Period: Overall Study
Arm/Group | Losartan
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Losartan
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Peak Eosinophil Count [Mean (Standard Deviation); unit: eosinophils per high power field] — Population: One subjects biopsies were not evaluated by research pathologist
  eosinophils per high power field
    Distal Peak Eosinophil Counts: number analyzed (Participants) | 5
    Distal Peak Eosinophil Counts | 108 (86)
    Proximal Peak Eosinophil Counts | 40 (37)
Pediatric EoE Symptom Score [Mean (Standard Deviation); unit: units on a scale] — Pediatric EoE Symptom score measures the frequency and severity of symptoms including nausea/vomiting, dysphagia, pain, and reflux. Scores range from 0 to 100. Higher scores indicate more frequent and/or severe symptoms. Population: Questionnaire not answered by one subject
  units on a scale
    number analyzed (Participants) | 5
    (all) | 28 (20)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants in Histologic Remission at 16 Weeks
Description: Percent of participants with peak eosinophil count < 15 eosinophils/high power field (remission) in distal and proximal esophagus
Time Frame: 16 weeks after treatment
Measure: Number; unit: percentage of participants
Arm/Group | Losartan
Number analyzed (Participants) | 6
percentage of participants
  Distal Remission | 17
  Proximal Remission | 17

2. Secondary Outcome: Change in Peak Eosinophil Count at 16 Weeks
Description: Mean change in peak eosinophil count from baseline
Time Frame: Baseline, 16 weeks after treatment
Measure: Mean (Standard Deviation); unit: eosinophils/high power field
Arm/Group | Losartan
Number analyzed (Participants) | 5
eosinophils/high power field
  Change in Distal Peak Count | -43 (107)
  Change in Proximal Peak Count | 3 (62)

3. Secondary Outcome: Change in Pediatric EoE Symptom Score at 16 Weeks
Description: The PEESS V2.0 questionnaire captures EoE-specific symptoms (dysphagia, GERD, nausea/vomiting, and pain) as reported by parents. The range for PEESS v2.0 scores is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms. Scores were obtained at baseline and 16 weeks. Change in score is defined as total score at 16 weeks minus total score at baseline.
Time Frame: Baseline, 16 weeks after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Losartan
Number analyzed (Participants) | 5
score on a scale | -11 (12)

ADVERSE EVENTS:
Time Frame: From consent to cessation of study which is approximately 24 weeks
Arm/Group | Losartan
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Food impaction (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hearing loss (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes